CLINICAL TRIAL: NCT07389161
Title: Uneven Nutrition and Life Style as IBD Triggers in Adolescents and Adults
Acronym: UNITA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Malmö University (Other); Lund University (Other); Linkoeping University (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-01188-01 UNITA
Record Dates: First submitted 2025-12-16; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Mb Crohn; Ulcerative Colitis (UC)
Keywords: Diet; Inflammatory bowel disease; Mb Crohn; Ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Sequential Assignment Prospective non-randomized intevention study where everyone serves as their own control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Intervention where every one serves as their own control
  Interventions: Dietary Supplement: Nordiet

INTERVENTIONS:
Dietary Supplement: Nordiet — Intervention with a Mediterranean like diet, the so called "Nordiet" during four weeks.

SUMMARY:
The aims of the study are 1. to determine the effect on dysbiosis, permeability and inflammatory activity after administration of a Mediterranean like diet (a Nordic equivalent, "Nordiet"), 2. to investigate life style related factors, such as exercise, psychosexual health and quality of life and their relation to the disease activity.

DETAILED DESCRIPTION:
The project aims, firstly, to map the quality of life and psychosexual health of young IBD patients (18-35 years), secondly, to investigate what treatment effect a changed diet can bring, and thirdly, to investigate whether physical activity and body composition can be related to disease activity.

The investigators want to use a natural food based on Mediterranean diet without artificial additives to evaluate the effect on the degree of disease activity through analysis of customary clinical parameters such as symptom picture and lab work including calprotectin (in stool samples) but mainly analysis of the gut microbiota and bacterial DNA in the blood as a marker for intestinal health.

Physical activity can be a possible treatment. By combining activity bracelets with analysis of autonomic balance (heart rate variability) and sleep quality, examinations of symptom burden and inflammatory activity, new valuable knowledge can be obtained.

Associations have been demonstrated between active IBD, depression, stress, fatigue, quality of life and sexual function in both women and men. It is therefore important to investigate psychosexual health and quality of life among young people with IBD and to also evaluate the effects of intervention through questionnaires and qualitative interviews.

ELIGIBILITY:
Inclusion Criteria:

* IBD, i.e., Mb Crohn or ulcerrative colitis
* Moderatively active disease (calprotectin 200-600)

Exclusion Criteria:

* Proctitis alone
* Inactive disease
* Severe flare up requiring in-patient care
* Planned change of treatment
* Antibiotic treatment during the last month
* Pregnancy
* Inability to understand Swedish
* Multimorbidity

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbial composition | Four weeks
  Gut microbiota will be analyzed at start and after four weeks. The health promoting efect of the diet will be estimated with analysis of the total bacterial genome down to species level. The bacterial composition will then be analyzed with regard to presence of beneficial or harmful bacteria. Based on the complexity of the micorbiota it is not possible to state any specific value that should be achieved.

SECONDARY OUTCOMES:
Disease activity | Four weeks
  Laboratory data:
  Calprotectin (mg/kg); lower level is better.
Disease activity | Four weeks
  Questionnaires:
  Harvey-Bradshaw Index (ulcerative colitis). Lower levels are in accordance with lower disease activity.
Disease activity | Four weeks
  Questionnaires:
  CDAI (Crohn's Disease Activity Index). Lower levels are in accordance with lower disease activity.

OTHER OUTCOMES:
Sleep quality | Four weeks.
  Activity bracelets will be used for measurements of sleep quality: This is based on a value that is a combination of time for sleep onset (minutes, shorter is better), the number of awakenings (fewer is better) and the amount of REM sleep during the night (minutes, more is better). A cut-off level is not appropriate. It is indvidual and must be based both on absolute outcome and relative change.

CONTACTS AND LOCATIONS:
Overall Officials: Vedrana Vejzovic, Associate professor, Study Director — Malmö University
Locations (1):
- Skåne University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data on group level can be shared upon request.
Supporting Information: Study Protocol, CSR
Time Frame: 2026 Feb 01 - 2029 Dec 31
Access Criteria: In order to establish research cooperation.